CLINICAL TRIAL: NCT01028339
Title: Mannitol Versus Hypertonic Saline to Treat Intracranial Hypertension After Severe Traumatic Brain Injury : a Comparative Study on the Effects on PtiO2 and Microdialysis Values
Brief Title: Mannitol vs HS to Treat ICHT After Severe TBI : Comparison on PtiO2 and Microdialysis Values
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients enrolled during 2 years
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Principal Investigator, BORET Henry, Médecin en chef, Direction Centrale du Service de Santé des Armées
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSH versus mannitol
Record Dates: First submitted 2009-12-03; First posted 2009-12-09 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; PtiO2; Cerebral microdialysis; Osmotherapy; hypertonic saline; mannitol
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Saline Solution, Hypertonic; Mannitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol (Active Comparator)
  Interventions: Drug: Mannitol
- Hypertonic saline (Experimental)
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: Hypertonic saline — 2 mL/kg of 7.5% hypertonic saline associated to hydroxyethyl starch
  Arms: Hypertonic saline
Drug: Mannitol — Mannitol
  Arms: Mannitol

SUMMARY:
The purpose of this study is to determine whether hypertonic saline is as much effective as mannitol to treat intracranial hypertension after traumatic brain injury and has at least the same effects on PtiO2 and cerebral metabolism studied through microdialysis.

DETAILED DESCRIPTION:
Mannitol is frequently used to treat intracranial hypertension after TBI. However, it can be deleterious, particularly through hyperdiuresis and risks of hypovolemia. It also needs volume compensation and induces logistical problem because of needs of high infused volume to achieve osmolar load and avoid hypotension. Finally, some recent studies tend to prove superiority of hypertonic saline versus mannitol on the prognosis of TBI. especially through modulation of inflammatory reactions mechanisms and apoptosis.

We would like to prove non inferiority of hypertonic saline versus mannitol after TBI to allow its large utilization, especially by field military doctors with specific logistical problems. For that, more than the single Intracranial Pressure, we want to study effects of HS vs mannitol not only on PtiO2 but also on cerebral microdialysis which gives informations on focal metabolism with profiles of ischemia, metabolic crisis, hyperglycolysis (possible reflect of neuronal restoration) and normality.

ELIGIBILITY:
Inclusion Criteria:

* Severe Traumatic brain injury monitored with ICP, PtiO2 and cerebral microdialysis
* And ICP> 20 mm Hg needing osmotherapy
* And approval of the next of kind

Exclusion Criteria:

* Bilateral fixed dilated pupils
* Contra-indication to multimodal neuromonitoring
* Previous CNS disease
* Contra-indication to HS (cardiac insufficiency,...)
* Natremia > 155 mmol/L or osmolarity > 320 mOsm/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Effects of HS versus mannitol on lactate/pyruvate ratio | 20 min, 40 min, H1, H2, H3 and H4

SECONDARY OUTCOMES:
Metabolic profile evaluated thanks to measure of lactate/pyruvate ratio and cerebral glucose | 20 min, 40 min, H1, H2, H3 and H4
Duration of PtiO2 > 15 mm Hg if PtiO2 was < 15 mm Hg before osmotherapy | 20 min, 40 min, H1, H2, H3 et H4
Duration of ICP<20 mm Hg after osmotherapy | 20 min, 40 min, H1, H2, H3 and H4
Interstitial osmolarity | 20 min, 40 min and H1
Necessity of a third line therapy (hypothermia, craniectomy, propofol/barbiturate coma | Day after osmotherapy
Length of stay | After leaving the unit
Mortality | 28th days
Glasgow outcome scale | 6th month

CONTACTS AND LOCATIONS:
Overall Officials: Henry BORET, MD, Principal Investigator — Direction Centrale du Service de Santé des Armées
Locations (1):
- HIA Sainte Anne, Toulon, France

REFERENCES:
- [Background] Vialet R, Albanese J, Thomachot L, Antonini F, Bourgouin A, Alliez B, Martin C. Isovolume hypertonic solutes (sodium chloride or mannitol) in the treatment of refractory posttraumatic intracranial hypertension: 2 mL/kg 7.5% saline is more effective than 2 mL/kg 20% mannitol. Crit Care Med. 2003 Jun;31(6):1683-7. doi: 10.1097/01.CCM.0000063268.91710.DF. PMID 12794404
- [Background] Sakowitz OW, Stover JF, Sarrafzadeh AS, Unterberg AW, Kiening KL. Effects of mannitol bolus administration on intracranial pressure, cerebral extracellular metabolites, and tissue oxygenation in severely head-injured patients. J Trauma. 2007 Feb;62(2):292-8. doi: 10.1097/01.ta.0000203560.03937.2d. PMID 17297315
- [Background] Soustiel JF, Vlodavsky E, Zaaroor M. Relative effects of mannitol and hypertonic saline on calpain activity, apoptosis and polymorphonuclear infiltration in traumatic focal brain injury. Brain Res. 2006 Jul 26;1101(1):136-44. doi: 10.1016/j.brainres.2006.05.045. Epub 2006 Jun 19. PMID 16787640